CLINICAL TRIAL: NCT00888758
Title: Randomized Comparison of Biolimus-Eluting and Everolimus-Eluting Stents With Optical Coherence Tomography Guided Stent Implantation in ST Elevation Myocardial Infarction.A 9-Month Angiographic and Optical Coherence Tomography Follow-up.
Brief Title: Comparison of Biolimus A9 and Everolimus Drug-Eluting Stents in Patients With ST Segment Elevation Myocardial Infarction
Acronym: ROBUST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Masaryk University (Other)
Responsible Party: Assoc. prof. Pavel Červinka, MD, PhD, FESC, FSCAI, Masaryk hospital and University of JEP Ústí nad Labem
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 06042006
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Heart Disease; Percutaneous Coronary Intervention
Keywords: Stents
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Device: biolimus A9
- 2 (Active Comparator)
  Interventions: Device: everolimus

INTERVENTIONS:
Device: biolimus A9 — 200 patients with STEMI will be treated using Biomatrix stent.
  Other Names: biolimus A9 eluting stent
  Arms: 1
Device: everolimus — 200 patients with STEMI will be treated with PROMUS DES.
  Other Names: everolimus eluting stent
  Arms: 2

SUMMARY:
The primary objective of this study is:

* comparison of a safety and effectiveness of third generation DES (biolimus A9 and everolimus) in patients with STEMI treated by primary PCI with OCT guidance. A rate of 9 month MACE (deaths, myocardial infarction, ischemia driven TLR) will be assessed in both groups.

The secondary outcomes are a comparison of (using OCT):

* number of uncovered stent struts
* number of malapposed stents struts
* in-stent neointimal volume
* in-segment assessment of vessel wall response to DES

DETAILED DESCRIPTION:
The aim of this multicenter, prospective, randomized trial with a core lab analysis is to assess the safety and effectiveness (at 9-month follow-up) of third generation DES (biolimus A9 and everolimus) in patients with evolving STEMI with the OCT guidance (to optimize a stent implantation) A serial OCT analysis will be performed to assess the number of either uncovered or malaposed stents strut and a degree of in-stent neointimal hyperplasia. Furthermore, the in-segment vessel wall response to DES implantation will also be analysed. The goal is to enroll 400 patients (200 in each group) with OCT guidance in 100 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Acute STEMI within 12 hours from symptoms onset
2. Native coronary disease with a lesion suitable for stenting
3. Vessel size in between 2.5-3.75mm
4. Patient is willing to provide written informed consent
5. Male or female patients between 18-85 years of age

Exclusion Criteria:

1. Significant left main disease
2. Killip class IV
3. Known allergy to aspirin and or clopidogrel/ticlopidine
4. Recent bleeding (<1month)
5. Patient in anticoagulant therapy
6. No suitable coronary anatomy for OCT scan (ostial lesion, very distal or large vessel />3.75mm in diameter/)
7. Pregnancy
8. Severe liver or renal disease (Cr>2.0)
9. Life expectancy < 1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-01 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
to compare a safety and effectiveness of third generation DES (biolimus A9 and everolimus) in patients with STEMI treated by primary PCI with OCT guidance with assessment of a MACE's at 9 month follow-up | 2 years

SECONDARY OUTCOMES:
number of uncovered stent struts | 2 years
number of malaposed stents struts | 2 years
in-stent neointimal volume | 2 years
in-segment assessment of vessel wall response to DES | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Cervinka, MD, PhD, Principal Investigator — Krajska zdravotni a.s., Masarzk hospital Usti nad Labem
Locations (1):
- Department of Cardiology, Masaryk hospital and University of JEP, Ústí nad Labem, Czechia